CLINICAL TRIAL: NCT02818699
Title: Body Fat Reducing Effect and Safety of Enzymatically Modified Isoquercitrin in Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2885
Record Dates: First submitted 2016-06-07; First posted 2016-06-30 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Capsule (Placebo Comparator): Participants assigned to this group will receive placebo capsules identical in appearance to EMIQ capsules.
  Interventions: Dietary Supplement: Placebo
- EMIQ Capsule (Experimental): Participants assigned to this group will receive EMIQ capsules identical in appearance to placebo capsules.
  Interventions: Dietary Supplement: EMIQ

INTERVENTIONS:
Dietary Supplement: Placebo — 280mg placebo capsule containing only maltodextrin, twice daily, one with breakfast, one with dinner, for 12 weeks
  Arms: Placebo Capsule
Dietary Supplement: EMIQ — 280mg placebo capsule containing 180 mg EMIQ and 100mg maltodextrin, twice daily, one with breakfast, one with dinner, for 12 weeks
  Arms: EMIQ Capsule

SUMMARY:
The purpose of this clinical study is to determine the effect and safety of long-term intake of enzymatically modified isoquercitrin (EMIQ), a natural plant product on body fat loss in obese and overweight individuals.

DETAILED DESCRIPTION:
This study is being conducted to assess the effect of supplementation with Enzymatically Modified Isoquercitrin (EMIQ) vs. placebo on measures of total body fat in overweight and obese adults. Participants will visit the HNRCA on 5 different dates.

Visit 1: Participants will receive materials and instruction for completing 24-hour dietary recalls to be completed by phone a week prior to the next visit.

Visit 2: Overnight fasted participants will arrive to the Human Nutrition Research Center on Aging (HNRCA). Vital signs, and EKG measure of heart rhythm, scrub weight and height will be obtained. Blood samples will be collected. Several baseline measurements will be performed during this visit including: lipid profile, insulin test, adiponectin, a urine dip stick, skinfold thickness and waist/hip circumference, resting metabolic rate (RMR), and DXA measure of total body fat. A three factor eating questionnaire, food craving questionnaire, and the Stanford 7-Day Physical Activity Recall (PAR) will be administered to assess volunteer's dietary inhibition, restraint, hunger, cravings and physical activity level. EMIQ and placebo capsules, compliance calendar, and instructions will be dispensed to participants by nursing staff.

Visit 3: Overnight fasted participants will arrive to HNRCA four weeks from the last visit. Participants will be asked to return their unused supplements as well as their compliance calendar. Vital signs, scrub weight and changes to volunteer health, medication and eligibility status will be assessed. Blood samples will be collected. A second EKG will be performed. The PAR will be administered. Before their next visit, participants will complete 3 24- hour dietary recalls by phone.

Visit 4: overnight fasted participants will arrive to HNRCA four weeks from the last visit. Participants will be asked to return their unused supplements as well as their compliance calendar. Vital signs, scrub weight and changes to volunteer health, medication and eligibility status will be assessed. Blood samples will be collected. The PAR will be administered. Before their next visit, participants will complete 3 24- hour dietary recalls by phone.

Visit 5: Overnight fasted participants will arrive to HNRCA four weeks from the last visit. Vital signs and scrub weight will be assessed. Blood samples will be collected. Final measurements will be taken during this visit including: routine health screening analysis, lipid profile, adiponectin, insulin test, a urine dip stick, liver and kidney function (SGOT, SGPT, BUN, creatinine, and calculated GFR), skin fold thickness, DXA, RMR and waist/hip circumference. A three factor eating questionnaire, food craving questionnaire, and the PAR will be administered to assess changes in volunteer's dietary inhibition, restraint, hunger, cravings and activity level throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-65 years.
* Premenopausal female with regular menstrual cycle or post-menopausal female with cessation of menstrual cycle for a minimum of 6 months.
* BMI in the range of 28.0-35.0
* Beck Depression Inventory Score less than 20.
* Fluency in spoken or written English.
* Willingness to be randomized to take EMIQ or placebo.
* Must weigh at least 164lbs

Exclusion Criteria:

* Any major illness or condition that may interfere with study outcomes at the discretion of the study physician.
* Diabetes Type I & Type II, or use of any pharmacological treatment for diabetes.
* Use of medications that interfere with energy metabolism
* Receiving hormone therapy growth hormone, testosterone, or estrogen with the exception of hormone contraceptives.
* GI diseases, conditions or medications known to influence GI absorption including active peptic ulcer disease or inflammatory bowel disease such as ulcerative colitis, Crohn's disease, celiac disease, chronic diarrhea or constipation.
* Undergone gastric bypass or other bariatric weight loss procedure.
* Lipid lowering medications such as: bile acid sequestrants (Cholestyramine, Colestipol, Colesevelam, etc.), cholesterol absorption inhibitors (Ezetimibe-Zetia), and fibrates (Gemfibrozil, Clofibrate, Fenofibrate, Triclor). Exceptions to this exclusion are 3-hydroxy-3-methyl-glutaryl-coenzyme A reductase (HMG-CoA reductase or Statins).
* On or planning to participate in a weight loss program.
* Weight loss or weight gain greater than 10 lbs in the past 6 months.
* History of eating disorders, anorexia, bulimia, or binge-eating in the past 5 years.
* Participation in any regular endurance exercise: running, biking or aerobics (except walking) greater than 2.5 hours per week, or resistance training greater than once per week.
* Regular use of acid lowering medications (greater than 3 times per week) such as antacids, proton pump inhibitors (PPIs), or H2 blockers.
* Unstable thyroid disease.
* Psychiatric disorders including schizophrenia, bipolar, major depression or psychosis.
* Antidepressant medication: selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase (MAO) inhibitors, or tricyclic antidepressants (TCAs).
* Cancer of any type (except for non-melanoma skin) in the past 5 years.
* Use of chemotherapeutic agents.
* Pregnancy, planning to become pregnant during the study period, or breastfeeding.
* Unwilling to use effective birth control during study.
* History of bilateral mastectomy with nodal dissection.
* Alcohol use, on average, greater than 3 servings per day, 20 servings per week (Serving size: 12oz beer, 4oz wine, 2oz hard liquor), or self-reported binge drinking.
* Uncontrolled hypertension (HTN) determined at the discretion of the study MD or registered nurse (RN). HTN medications allowed in the study: angiotensin converting enzyme (ACE) inhibitors, calcium channel blockers, and diuretics.
* Medications for chronic obstructive pulmonary disease (COPD) or kidney disease.
* α-adrenergic or β-adrenergic blockers (oral or ocular) and diuretics.
* Renal or chronic kidney disease due to any condition, renovascular disease, or dialysis.
* Chronic liver disease such as hepatitis B, hepatitis C, or cirrhosis.
* Cardiovascular disease including: myocardial infarction, cerebrovascular disease (CVA), coronary artery bypass graft, stenosis greater than 50%, angina, coronary artery disease (CAD), congestive heart failure (CHF),peripheral vascular disease (PVD) or dysautonomia.
* History of autoimmune diseases such as rheumatoid arthritis, lupus, multiple sclerosis, vitiligo, or psoriasis.
* HIV or AIDS based on self-report.
* Steroid use with the exception of over-the-counter topical and nasal steroids such as Flonase.
* Allergy medication or regular antihistamine use.
* Seizure disorders. Acceptable if managed with medication and free of seizure activity for 5 years.
* Smoking or the use of nicotine replacement products in the past 6 months.
* Use of dietary supplements containing vitamins (except Calcium and Vitamin D), minerals, herbal or plant-based preparations, fish oil or homeopathic remedies during study participation unless willing to discontinue prior to enrollment.
* Current participation in another research study.
* Non-English speaking.
* No social security number.
* Participation in another research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Body Fat | Change from baseline at 12 weeks
  Whole body fat measured by both dual-energy X-ray absorptiometry (DXA) and skin fold thickness

SECONDARY OUTCOMES:
Anthropomorphic Measure I | Change from baseline after 4 weeks, after 8 weeks and after 12 weeks
  Body weight
Anthropomorphic Measure II | Change from baseline at 12 weeks.
  Waist/Hip circumference
Metabolic Syndrome Measure I | Change from baseline at 12 weeks.
  Triglycerides
Metabolic Syndrome Measure II | Change from baseline at 12 weeks.
  Total Cholesterol
Metabolic Syndrome Measure III | Change from baseline at 12 weeks.
  HDL
Metabolic Syndrome Measure IV | Change from baseline at 12 weeks.
  LDL
Metabolic Syndrome Measure V | Change from baseline at 12 weeks.
  Insulin
Metabolic Syndrome Measure VI | Change from baseline at 12 weeks.
  Adiponectin.
Total protein | Change from baseline at 12 weeks.
  Total protein measured in urine.
Glucose | Change from baseline at 12 weeks.
  Glucose measured in urine.
Urobilinogen | Change from baseline at 12 weeks.
  Urobilinogen measured in urine.
Bilirubin | Change from baseline at 12 weeks.
  Bilirubin measured in urine.
Urine acidity | Change from baseline at 12 weeks.
  Hydrogen ion concentration (pH) measured in urine.
Ketones | Change from baseline at 12 weeks.
  Ketones measured in urine.
Occult Blood | Change from baseline at 12 weeks.
  Occult blood count measured in urine.
Resting Metabolic Rate | Change from baseline at 12 weeks.
  Used to determine rate of calories burned per day.
Nutritional Intake | Measures taken at baseline, week 6 and week 12.
  Nutritional intake measures assessed via 3 sets of 3 24-hour dietary recalls by phone.
Three Factor Eating Questionnaire | Changes from baseline after 12 weeks.
  Dietary restraint, disinhibition and hunger measured by Three Factor Eating questionnaire.
Food Cravings | Changes from baseline after 12 weeks.
  Changes in food cravings assessed by Food Cravings-Trait questionnaire
Physical Activity | Changes from baseline at 4, 6 8 and 12 weeks.
  Physical activity tracked and measured with the Stanford 7-Day Physical Activity Recall questionnaire.
Mental Health | Change from screening to end of study (approximately 14 weeks)
  Depression assessed by the Beck Depression Inventory.
Heart Health | Change from baseline at 4 weeks.
  Electrocardiogram (EKG) will be used to assess changes to heart rhythm.
Liver Health Marker I | Change from baseline after 4 weeks, after 8 weeks and after 12 weeks.
  Serum glutamic pyruvic transaminase (SGPT)
Liver Health Marker II | Change from baseline after 4 weeks, after 8 weeks and after 12 weeks.
  Serum glutamic oxaloacetic transaminase (SGOT).
Kidney Health Measure I | Change from baseline after 4 weeks, after 8 weeks and after 12 weeks.
  Blood urea nitrogen (BUN).
Kidney Health Measure II | Change from baseline after 4 weeks, after 8 weeks and after 12 weeks.
  Creatinine concentration.
Kidney Health Measure III | Change from baseline after 4 weeks, after 8 weeks and after 12 weeks.
  Glomerular filtration rate (GFR).

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Meydani, DVM, PhD, Principal Investigator — USDA Human Nutrition Research Center on Aging
Locations (1):
- Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT02818699/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT02818699/SAP_001.pdf